CLINICAL TRIAL: NCT00935012
Title: Open-Label Safety And Efficacy Evaluation Of Fx-1006a In Patients With V122i Or Wild-Type Transthyretin (TTR) Amyloid Cardiomyopathy
Brief Title: Safety And Efficacy Evaluation Of Fx-1006a In Patients With V122i Or Wild-Type Transthyretin (TTR) Amyloid Cardiomyopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX1B-303; B3461026 (Other: Alias Study Number)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: ATTR-CM; TTR-CM
Keywords: TTR, ATTR, cardiomyopathy, amyloidosis, tafamidis
MeSH Terms: conditions — Cardiomyopathies; Amyloidosis | interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label (Experimental)
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — Once daily 20 mg oral tafamidis (soft gelatin capsule)

SUMMARY:
Open-label Safety and Efficacy Evaluation of Fx-1006a in Patients with V122i Or Wild-type Transthyretin (ttr) Amyloid Cardiomyopathy.

Patients who successfully complete Fx1B-201 will report to the clinical unit on Day 0 to sign the informed consent form and determine eligibility for Protocol Fx1B-303. In addition, on Day 0, patients will have their entrance criteria reviewed, and medical histories and demographic characteristics obtained.

The physical examination (including weight and vital signs) and the relevant end of study clinical laboratory tests (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, gamma glutamyl transferase, creatinine, total bilirubin, international normalized ratio, troponin I, troponin T, and amino-terminal B-type natriuretic peptide) from Protocol Fx1B-201 will be used for Protocol Fx1B-303. If more than 30 days has elapsed between the final study visit of Protocol Fx1B-201 and Day 0 of Protocol Fx1B-303, an abbreviated physical examination (including weight and vital signs) and clinical laboratory assessments must be performed on Day 0.

Eligible patients will begin once-daily dosing with 20 mg Fx-1006A at home on Day 1 (i.e., first dose) and will return to the clinical unit for study visits every 6 months.

Adverse events (AEs) and concomitant medication use will be collected at each 6-month visit to the clinical unit. Blood draws for clinical safety laboratory tests and abbreviated physical examinations (including weight and vital signs) will also be performed at each 6-month clinic visit. ECGs will be performed every 12 months on an annual basis. A telephone call will be made at 3-month intervals between clinic visits to assess safety and use of concomitant medications.

For the evaluation of efficacy, the Patient Global Assessment, NYHA classification, KCCQ, 6-minute walk test, and efficacy-related clinical laboratory tests (serum levels of troponin T, troponin I, and NT-pro-BNP) will be determined every 6 months. In addition, echocardiograms will be performed every 12 months on an annual basis.

An end of study visit including all safety and efficacy assessments will occur upon patient completion of the study, premature withdrawal (for any reason), or in the event of program discontinuation by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patient successfully completed Protocol Fx1B-201.
* If female; patient is post menopausal. If male, female partner is post-menopausal. If female is of child bearing potential, willing to use acceptable method of birth control up to 3 months after last dose (included female partners of male participants).
* Patient is willing to comply with protocol.

Exclusion Criteria:

* Patient did not successfully complete Fx1B-201.
* Chronic use of NSAIDS.
* Patient has a clinically significant medication condition that increases risk of study participation.
* Patient has received heart or liver transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Emory University School of Medicine, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Cardiovascular Research Laboratory for the Elderly (CCRLE), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FX1B-303&StudyName=Safety%20And%20Efficacy%20Evaluation%20Of%20Fx-1006a%20In%20Patients%20With%20V122i%20Or%20Wild-Type%20Transthyretin%20%28TTR%29%20Amyloid%20Cardiomyopathy%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with transthyretin amyloid cardiomyopathy (TTR-CM/ATTR-CM), who had not undergone liver or heart transplantation and who had completed previous study Fx1B-201 (NCT00694161) were eligible to enter this current study Fx1B-303 (NCT00935012).
Pre-assignment Details: In this study, participants continued on same dose they had received in initial study. Data for time points from Baseline to Month 12 are from study Fx1B-201, while data for time points after Month 12 are from study Fx1B-303.
Groups:
- Tafamidis 20 mg: Participants received tafamidis 20 milligram (mg) soft gelatin capsule orally once daily for up to 10 years from the date of enrollment in this study (Fx1B-303) or until they had an access to tafamidis for TTR-CM via prescription, upon regulatory approval in respective countries.
Period: Overall Study
Arm/Group | Tafamidis 20 mg
Started | 31
Completed | 2
Not Completed | 29
Not completed — Death | 19
Not completed — Withdrawal by Subject | 3
Not completed — Other | 5
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure.
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
  Afro-caribbean | 1
  African American | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Categories of Patient Global Assessment (PGA) for Follow-up Visit: Month 12
Description: Participants overall quality of life was measured by PGA. At follow-up visit, participants were asked, "How do you feel today as compared to when we talked with you at your last clinic visit for this study?" and participants responded to any of the following: markedly improved, moderately improved, mildly improved, unchanged, mildly worsened, moderately worsened or markedly worsened.
Time Frame: Month 12
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
percentage of participants
  Markedly Improved | 0 [0.0 to 11.2]
  Moderately Improved | 16.1 [5.5 to 33.7]
  Mildly Improved | 9.7 [2.0 to 25.8]
  Unchanged | 51.6 [33.1 to 69.8]
  Mildly Worsened | 12.9 [3.6 to 29.8]
  Moderately Worsened | 9.7 [2.0 to 25.8]
  Markedly Worsened | 0 [0.0 to 11.2]

2. Primary Outcome: Percentage of Participants With Categories of Patient Global Assessment (PGA) for Follow-up Visit: Month 60
Description: as for outcome 1
Time Frame: Month 60
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
percentage of participants
  Markedly Improved | 0 [0.0 to 26.5]
  Moderately Improved | 8.3 [0.2 to 38.5]
  Mildly Improved | 8.3 [0.2 to 38.5]
  Unchanged | 50.0 [21.1 to 78.9]
  Mildly Worsened | 16.7 [2.1 to 48.4]
  Moderately Worsened | 16.7 [2.1 to 48.4]
  Markedly Worsened | 0 [0.0 to 26.5]

3. Primary Outcome: Number of Participants Classified on the Basis of New York Heart Association (NYHA) Classification at Baseline
Description: NYHA classified participants in 4 classes. Class I included participants with cardiac disease without limitations of physical activity. Ordinary physical activity did not cause undue fatigue, palpitation, dyspnea, or anginal pain. Class II included participants with cardiac disease with slight limitation of physical activity. They were comfortable at rest. Ordinary physical activity resulted in fatigue, palpitation, dyspnea, or anginal pain. Class III included participants with cardiac disease with marked limitation of physical activity. They were comfortable at rest. Less than ordinary physical activity caused fatigue, palpitation, dyspnea, or anginal pain. Class IV included participants with cardiac disease with the inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome might be present even at rest. If any physical activity was undertaken, discomfort was increased.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants
  CLASS I | 4
  CLASS II | 26
  CLASS III | 1
  CLASS IV | 0

4. Primary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Classification at Month 12
Description: NYHA classified participants in 4 classes: Class I: cardiac disease without limitations of physical activity. Ordinary physical activity caused no undue fatigue, palpitation, dyspnea or angina pain. Class II: cardiac disease with slight limitation of physical activity, comfortable at rest. Ordinary physical activity resulted in fatigue, palpitation, dyspnea or angina pain. Class III: cardiac disease with marked limitation of physical activity, comfortable at rest. Less than ordinary physical activity caused fatigue, palpitation, dyspnea or angina pain. Class IV: cardiac disease with inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or angina syndrome might be present even at rest. If any physical activity was undertaken, discomfort was increased. Participants with change from baseline were classified as improved (shifted from higher to lower class), unchanged (no change in class) or worsened (shifted from lower to higher class).
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants
  Worsened | 7
  Unchanged | 20
  Improved | 4

5. Primary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Classification at Month 60
Description: as for outcome 4
Time Frame: Baseline, Month 60
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 12
Participants
  Worsened | 8
  Unchanged | 3
  Improved | 1

6. Primary Outcome: Change From Baseline in Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 12
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. In this outcome measure, the total distance that a participant could walk in 6 minutes was evaluated.
Time Frame: Baseline, Month 12
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure. "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure. "Number analyzed" =participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 30
meters
  Baseline | 363.7 (130.80)
  Change at Month 12: number analyzed (Participants) | 28
  Change at Month 12 | -11.2 (76.39)

7. Primary Outcome: Change From Baseline in Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 60
Description: as for outcome 6
Time Frame: Baseline, Month 60
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 8
meters | -121.4 (145.82)

8. Primary Outcome: Number of Participants Categorized Based on Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 12
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. In this outcome measure, participants were categorized based on the total distance walked as Level 1 = total distance walked less than (<) 300 meter; Level 2 = total distance walked between 300 to 374.9 meter; Level 3 = total distance walked between 375 to 449.9 meter; Level 4 = total distance walked greater than or equal to (>=) 450 meter.
Time Frame: Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 28
Participants
  Level 1 | 8
  Level 2 | 7
  Level 3 | 7
  Level 4 | 6

9. Primary Outcome: Number of Participants Categorized Based on Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 60
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. In this outcome measure, participants were categorized based on the total distance walked as Level 1 = total distance walked < 300 meter; Level 2 = total distance walked between 300 to 374.9 meter; Level 3 = total distance walked between 375 to 449.9 meter; Level 4 = total distance walked >=450 meter.
Time Frame: Month 60
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 8
Participants
  Level 1 | 4
  Level 2 | 3
  Level 3 | 0
  Level 4 | 1

10. Primary Outcome: Change From Baseline in Dyspnea and Fatigue Scores During 6 Minute Walk Test (6MWT) at Month 12
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. Dyspnea: participants were asked to rate the difficulty of their breathing, pre-walk and post-walk at each visit, on a scale of range 0 (no breathlessness at all) to 10 (maximum breathlessness). Higher scores indicated more severity. Fatigue: participants were asked to rate the how tired they felt, pre-walk and post-walk at each visit, on a scale of range 0 (not at all) to 10 (maximal) Higher scores indicated more fatigue. At each visit, scores for pre-walk test, post-walk test and within visit difference (difference from post-walk to pre-walk) were evaluated. Change from baseline was calculated for each pre-walk test, post-walk test and within visit difference at Month 12.
Time Frame: Baseline, Month 12
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure. "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure. "Number analyzed"=participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 28
units on a scale
  Dyspnea: Baseline, Pre walk | 0.6 (0.72)
  Dyspnea: Baseline, Post walk | 2.5 (1.94)
  Dyspnea: Baseline, Within Visit Difference | 1.9 (1.94)
  Dyspnea: Change at Month 12, Pre walk: number analyzed (Participants) | 26
  Dyspnea: Change at Month 12, Pre walk | 0.6 (1.61)
  Dyspnea: Change at Month 12, Post walk: number analyzed (Participants) | 26
  Dyspnea: Change at Month 12, Post walk | 1.2 (1.60)
  Dyspnea:Change at Month 12,Within Visit Difference: number analyzed (Participants) | 26
  Dyspnea:Change at Month 12,Within Visit Difference | 0.6 (1.70)
  Fatigue: Baseline, Pre-walk | 0.9 (1.27)
  Fatigue: Baseline, Post-walk | 2.4 (2.06)
  Fatigue: Baseline, Within Visit Difference | 1.4 (2.51)
  Fatigue: Change at Month 12, Pre Walk: number analyzed (Participants) | 26
  Fatigue: Change at Month 12, Pre Walk | 0.5 (2.20)
  Fatigue: Change at Month 12, Post-Walk: number analyzed (Participants) | 26
  Fatigue: Change at Month 12, Post-Walk | 0.9 (1.98)
  Fatigue:Change at Month 12,Within Visit Difference: number analyzed (Participants) | 26
  Fatigue:Change at Month 12,Within Visit Difference | 0.4 (2.20)

11. Primary Outcome: Change From Baseline in Dyspnea and Fatigue Scores During 6 Minute Walk Test (6MWT) at Month 60
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. Dyspnea: participants were asked to rate the difficulty of their breathing, pre-walk and post-walk at each visit, on a scale of range 0 (no breathlessness at all) to 10 (maximum breathlessness). Higher scores indicated more severity. Fatigue: participants were asked to rate the how tired they felt, pre-walk and post-walk at each visit, on a scale of range 0 (not at all) to 10 (maximal) Higher scores indicated more fatigue. At each visit, scores for pre-walk test, post-walk test and within visit difference (difference from post-walk to pre-walk) were evaluated. Change from baseline was calculated for each pre-walk test, post-walk test and within visit difference at Month 60.
Time Frame: Baseline, Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 8
units on a scale
  Dyspnea: Change at Month 60, Pre walk | 0.8 (1.41)
  Dyspnea: Change at Month 60, Post walk | 0.8 (1.60)
  Dyspnea:Change at Month 60,Within Visit Difference | 0.1 (1.94)
  Fatigue: Change at Month 60, Pre walk | 0.1 (0.35)
  Fatigue: Change at Month 60, Post walk | 0.4 (1.51)
  Fatigue:Change at Month 60,Within Visit Difference | 0.3 (1.49)

12. Primary Outcome: Number of Participants Categorized on Basis of Change From Baseline in Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 12
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. In this outcome measure, participants on basis of change from baseline in total distance walked were categorized as worsened, unchanged or improved. If distance walked at a visit was greater than distance walked at baseline, then categorized as 'improved'. If distance walked at a visit was equal to distance walked at baseline, then categorized as 'unchanged'. If distance walked at a visit was less than distance walked at baseline, then categorized as 'worsened'.
Time Frame: Baseline, Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 28
Participants
  Worsened | 7
  Unchanged | 16
  Improved | 5

13. Primary Outcome: Number of Participants Categorized on Basis of Change From Baseline in Total Distance Walked During 6 Minute Walk Test (6MWT) at Month 60
Description: as for outcome 12
Time Frame: Baseline, Month 60
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 8
Participants
  Worsened | 5
  Unchanged | 3
  Improved | 0

14. Primary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Summary Score at Month 12
Description: KCCQ is a 23-item participant-completed questionnaire that assesses health status and health-related quality of life in participants with heart failure. Eight domain scores were calculated for the KCCQ: physical limitation, social limitation, quality of life, self-efficacy, symptom stability, symptom frequency, symptom burden, and total symptoms (calculated as the mean of symptom frequency and symptom burden scores). Two summary scores were calculated: clinical summary (calculated as mean of physical limitation and total symptom scores) and overall summary (calculated as mean of physical limitation, social limitation, total symptoms, and quality of life scores). Each domain and both summary scores were scaled to range from 0 (worse health status) to 100 (best health status); higher scores represented better health status.
Time Frame: Baseline, Month 12
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure. "Number analyzed" =participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
units on a scale
  Overall Summary Score: Baseline | 72.21 (18.974)
  Overall Summary Score: Change at Month 12: number analyzed (Participants) | 30
  Overall Summary Score: Change at Month 12 | -4.54 (12.724)
  Clinical Summary Score: Baseline | 74.79 (19.296)
  Clinical Summary Score: Change at Month 12: number analyzed (Participants) | 30
  Clinical Summary Score: Change at Month 12 | -5.60 (13.792)

15. Primary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Summary Score at Month 60
Description: as for outcome 14
Time Frame: Baseline, Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 11
units on a scale
  Overall Summary Score: Change at Month 60 | -12.93 (29.306)
  Clinical Summary Score: Change at Month 60 | -18.12 (29.432)

16. Primary Outcome: Change From Baseline in Troponin I and Troponin T Serum Levels at Month 12
Description: Troponin I and troponin T are the cardiac markers. Troponin I and troponin T are part of the troponin complex, where troponin I is bound to actin in thin myofilaments and troponin T is bound to tropomyosin. Higher level of these markers is indicative of heart damage.
Time Frame: Baseline, Month 12
Population: Safety analysis population included all participants who were enrolled in this study and who had taken at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
nanogram per milliliter
  Troponin I: Baseline | 0.132 (0.0627)
  Troponin I: Change at Month 12 | 0.016 (0.0652)
  Troponin T: Baseline | 0.0448 (0.03402)
  Troponin T: Change at Month 12 | 0.0110 (0.02239)

17. Primary Outcome: Change From Baseline in Troponin I and Troponin T Serum Levels at Month 60
Description: as for outcome 16
Time Frame: Baseline, Month 60
Population: Safety analysis population included all participants who were enrolled in this study and who had taken at least 1 dose of study medication. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure. "Number analyzed" =participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 11
nanogram per milliliter
  Troponin T: Change at Month 60 | 0.026 (0.0937)
  Troponin I: Change at Month 60: number analyzed (Participants) | 10
  Troponin I: Change at Month 60 | 0.0810 (0.17779)

18. Primary Outcome: Change From Baseline in Amino-Terminal B-type Natriuretic Peptide (NT-proBNP) Serum Level at Month 12
Description: NT-proBNP is biomarker of cardiac stress (myocardial necrosis and increased filling pressures/ left ventricular [LV] wall stress).
Time Frame: Baseline, Month 12
Population: Safety analysis population included all participants who were enrolled in this study and who had taken at least 1 dose of study medication. "Number analyzed" =participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
nanogram per milliliter
  Baseline | 4526.1 (3814.21)
  Change at Month 12: number analyzed (Participants) | 30
  Change at Month 12 | 818.3 (3133.86)

19. Primary Outcome: Change From Baseline in Serum Levels of Amino-Terminal B-type Natriuretic Peptide (NT-proBNP) at Month 60
Description: NT-proBNP is biomarker of cardiac stress (myocardial necrosis and increased filling pressures/ LV wall stress).
Time Frame: Baseline, Month 60
Population: Safety analysis population consisted of all participants who were enrolled in this study and who had taken at least one dose of study medication. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 11
nanogram per milliliter | 5127.6 (10598.94)

20. Secondary Outcome: Percentage of Participants With Categories of Patient Global Assessment (PGA) for Follow-up Visit: Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126 and 132
Description: Participants overall quality of life was measured by PGA. At each follow-up visit, participants were asked, "How do you feel today as compared to when we talked with you at your last clinic visit for this study?" and participants responded to any of the following: markedly improved, moderately improved, mildly improved, unchanged, mildly worsened, moderately worsened or markedly worsened.
Time Frame: Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126, 132
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
percentage of participants
  Month 6: Markedly Improved | 9.7 [2.0 to 25.8]
  Month 6: Moderately Improved | 3.2 [0.1 to 16.7]
  Month 6: Mildly Improved | 9.7 [2.0 to 25.8]
  Month 6: Unchanged | 51.6 [33.1 to 69.8]
  Month 6: Mildly Worsened | 25.8 [11.9 to 44.6]
  Month 6: Moderately Worsened | 0 [0.0 to 11.2]
  Month 6: Markedly Worsened | 0 [0.0 to 11.2]
  Month 18: Markedly Improved: number analyzed (Participants) | 28
  Month 18: Markedly Improved | 7.1 [0.9 to 23.5]
  Month 18: Moderately Improved: number analyzed (Participants) | 28
  Month 18: Moderately Improved | 10.7 [2.3 to 28.2]
  Month 18: Mildly Improved: number analyzed (Participants) | 28
  Month 18: Mildly Improved | 17.9 [6.1 to 36.9]
  Month 18: Unchanged: number analyzed (Participants) | 28
  Month 18: Unchanged | 25.0 [10.7 to 44.9]
  Month 18: Mildly Worsened: number analyzed (Participants) | 28
  Month 18: Mildly Worsened | 17.9 [6.1 to 36.9]
  Month 18: Moderately Worsened: number analyzed (Participants) | 28
  Month 18: Moderately Worsened | 10.7 [2.3 to 28.2]
  Month 18: Markedly Worsened: number analyzed (Participants) | 28
  Month 18: Markedly Worsened | 10.7 [2.3 to 28.2]
  Month 24: Markedly Improved: number analyzed (Participants) | 22
  Month 24: Markedly Improved | 9.1 [1.1 to 29.2]
  Month 24: Moderately Improved: number analyzed (Participants) | 22
  Month 24: Moderately Improved | 18.2 [5.2 to 40.3]
  Month 24: Mildly Improved: number analyzed (Participants) | 22
  Month 24: Mildly Improved | 13.6 [2.9 to 34.9]
  Month 24: Unchanged: number analyzed (Participants) | 22
  Month 24: Unchanged | 27.3 [10.7 to 50.2]
  Month 24: Mildly Worsened: number analyzed (Participants) | 22
  Month 24: Mildly Worsened | 22.7 [7.8 to 45.4]
  Month 24: Moderately Worsened: number analyzed (Participants) | 22
  Month 24: Moderately Worsened | 4.5 [0.1 to 22.8]
  Month 24: Markedly Worsened: number analyzed (Participants) | 22
  Month 24: Markedly Worsened | 4.5 [0.1 to 22.8]
  Month 30: Markedly Improved: number analyzed (Participants) | 20
  Month 30: Markedly Improved | 0 [0.0 to 16.8]
  Month 30: Moderately Improved: number analyzed (Participants) | 20
  Month 30: Moderately Improved | 10.0 [1.2 to 31.7]
  Month 30: Mildly Improved: number analyzed (Participants) | 20
  Month 30: Mildly Improved | 5.0 [0.1 to 24.9]
  Month 30: Unchanged: number analyzed (Participants) | 20
  Month 30: Unchanged | 40.0 [19.1 to 63.9]
  Month 30: Mildly Worsened: number analyzed (Participants) | 20
  Month 30: Mildly Worsened | 25.0 [8.7 to 49.1]
  Month 30: Moderately Worsened: number analyzed (Participants) | 20
  Month 30: Moderately Worsened | 20.0 [5.7 to 43.7]
  Month 30: Markedly Worsened: number analyzed (Participants) | 20
  Month 30: Markedly Worsened | 0 [0.0 to 16.8]
  Month 36: Markedly Improved: number analyzed (Participants) | 19
  Month 36: Markedly Improved | 0 [0.0 to 17.6]
  Month 36: Moderately Improved: number analyzed (Participants) | 19
  Month 36: Moderately Improved | 0 [0.0 to 17.6]
  Month 36: Mildly Improved: number analyzed (Participants) | 19
  Month 36: Mildly Improved | 5.3 [0.1 to 26.0]
  Month 36: Unchanged: number analyzed (Participants) | 19
  Month 36: Unchanged | 47.4 [24.4 to 71.1]
  Month 36: Mildly Worsened: number analyzed (Participants) | 19
  Month 36: Mildly Worsened | 26.3 [9.1 to 51.2]
  Month 36: Moderately Worsened: number analyzed (Participants) | 19
  Month 36: Moderately Worsened | 21.1 [6.1 to 45.6]
  Month 36: Markedly Worsened: number analyzed (Participants) | 19
  Month 36: Markedly Worsened | 0 [0.0 to 17.6]
  Month 42: Markedly Improved: number analyzed (Participants) | 17
  Month 42: Markedly Improved | 0 [0.0 to 19.5]
  Month 42: Moderately Improved: number analyzed (Participants) | 17
  Month 42: Moderately Improved | 0 [0.0 to 19.5]
  Month 42: Mildly Improved: number analyzed (Participants) | 17
  Month 42: Mildly Improved | 0 [0.0 to 19.5]
  Month 42: Unchanged: number analyzed (Participants) | 17
  Month 42: Unchanged | 29.4 [10.3 to 56.0]
  Month 42: Mildly Worsened: number analyzed (Participants) | 17
  Month 42: Mildly Worsened | 35.3 [14.2 to 61.7]
  Month 42: Moderately Worsened: number analyzed (Participants) | 17
  Month 42: Moderately Worsened | 11.8 [1.5 to 36.4]
  Month 42: Markedly Worsened: number analyzed (Participants) | 17
  Month 42: Markedly Worsened | 23.5 [6.8 to 49.9]
  Month 48: Markedly Improved: number analyzed (Participants) | 13
  Month 48: Markedly Improved | 0 [0.0 to 24.7]
  Month 48: Moderately Improved: number analyzed (Participants) | 13
  Month 48: Moderately Improved | 0 [0.0 to 24.7]
  Month 48: Mildly Improved: number analyzed (Participants) | 13
  Month 48: Mildly Improved | 23.1 [5.0 to 53.8]
  Month 48: Unchanged: number analyzed (Participants) | 13
  Month 48: Unchanged | 53.8 [25.1 to 80.8]
  Month 48: Mildly Worsened: number analyzed (Participants) | 13
  Month 48: Mildly Worsened | 15.4 [1.9 to 45.4]
  Month 48: Moderately Worsened: number analyzed (Participants) | 13
  Month 48: Moderately Worsened | 7.7 [0.2 to 36.0]
  Month 48: Markedly Worsened: number analyzed (Participants) | 13
  Month 48: Markedly Worsened | 0 [0.0 to 24.7]
  Month 54: Markedly Improved: number analyzed (Participants) | 13
  Month 54: Markedly Improved | 0 [0.0 to 24.7]
  Month 54: Moderately Improved: number analyzed (Participants) | 13
  Month 54: Moderately Improved | 7.7 [0.2 to 36.0]
  Month 54: Mildly Improved: number analyzed (Participants) | 13
  Month 54: Mildly Improved | 0 [0.0 to 24.7]
  Month 54: Unchanged: number analyzed (Participants) | 13
  Month 54: Unchanged | 61.5 [31.6 to 86.1]
  Month 54: Mildly Worsened: number analyzed (Participants) | 13
  Month 54: Mildly Worsened | 23.1 [5.0 to 53.8]
  Month 54: Moderately Worsened: number analyzed (Participants) | 13
  Month 54: Moderately Worsened | 7.7 [0.2 to 36.0]
  Month 54: Markedly Worsened: number analyzed (Participants) | 13
  Month 54: Markedly Worsened | 0 [0.0 to 24.7]
  Month 66: Markedly Improved: number analyzed (Participants) | 6
  Month 66: Markedly Improved | 16.7 [0.4 to 64.1]
  Month 66: Moderately Improved: number analyzed (Participants) | 6
  Month 66: Moderately Improved | 0 [0.0 to 45.9]
  Month 66: Mildly Improved: number analyzed (Participants) | 6
  Month 66: Mildly Improved | 0 [0.0 to 45.9]
  Month 66: Unchanged: number analyzed (Participants) | 6
  Month 66: Unchanged | 50.0 [11.8 to 88.2]
  Month 66: Mildly Worsened: number analyzed (Participants) | 6
  Month 66: Mildly Worsened | 0 [0.0 to 45.9]
  Month 66: Moderately Worsened: number analyzed (Participants) | 6
  Month 66: Moderately Worsened | 33.3 [4.3 to 77.7]
  Month 66: Markedly Worsened: number analyzed (Participants) | 6
  Month 66: Markedly Worsened | 0 [0.0 to 45.9]
  Month 72: Markedly Improved: number analyzed (Participants) | 7
  Month 72: Markedly Improved | 0 [0.0 to 41.0]
  Month 72: Moderately Improved: number analyzed (Participants) | 7
  Month 72: Moderately Improved | 0 [0.0 to 41.0]
  Month 72: Mildly Improved: number analyzed (Participants) | 7
  Month 72: Mildly Improved | 0 [0.0 to 41.0]
  Month 72: Unchanged: number analyzed (Participants) | 7
  Month 72: Unchanged | 71.4 [29.0 to 96.3]
  Month 72: Mildly Worsened: number analyzed (Participants) | 7
  Month 72: Mildly Worsened | 28.6 [3.7 to 71.0]
  Month 72: Moderately Worsened: number analyzed (Participants) | 7
  Month 72: Moderately Worsened | 0 [0.0 to 41.0]
  Month 72: Markedly Worsened: number analyzed (Participants) | 7
  Month 72: Markedly Worsened | 0 [0.0 to 41.0]
  Month 78: Markedly Improved: number analyzed (Participants) | 7
  Month 78: Markedly Improved | 14.3 [0.4 to 57.9]
  Month 78: Moderately Improved: number analyzed (Participants) | 7
  Month 78: Moderately Improved | 0 [0.0 to 41.0]
  Month 78: Mildly Improved: number analyzed (Participants) | 7
  Month 78: Mildly Improved | 0 [0.0 to 41.0]
  Month 78: Unchanged: number analyzed (Participants) | 7
  Month 78: Unchanged | 28.6 [3.7 to 71.0]
  Month 78: Mildly Worsened: number analyzed (Participants) | 7
  Month 78: Mildly Worsened | 28.6 [3.7 to 71.0]
  Month 78: Moderately Worsened: number analyzed (Participants) | 7
  Month 78: Moderately Worsened | 28.6 [3.7 to 71.0]
  Month 78: Markedly Worsened: number analyzed (Participants) | 7
  Month 78: Markedly Worsened | 0 [0.0 to 41.0]
  Month 84: Markedly Improved: number analyzed (Participants) | 6
  Month 84: Markedly Improved | 16.7 [0.4 to 64.1]
  Month 84: Moderately Improved: number analyzed (Participants) | 6
  Month 84: Moderately Improved | 0 [0.0 to 45.9]
  Month 84: Mildly Improved: number analyzed (Participants) | 6
  Month 84: Mildly Improved | 0 [0.0 to 45.9]
  Month 84: Unchanged: number analyzed (Participants) | 6
  Month 84: Unchanged | 33.3 [4.3 to 77.7]
  Month 84: Mildly Worsened: number analyzed (Participants) | 6
  Month 84: Mildly Worsened | 16.7 [0.4 to 64.1]
  Month 84: Moderately Worsened: number analyzed (Participants) | 6
  Month 84: Moderately Worsened | 16.7 [0.4 to 64.1]
  Month 84: Markedly Worsened: number analyzed (Participants) | 6
  Month 84: Markedly Worsened | 16.7 [0.4 to 64.1]
  Month 90: Markedly Improved: number analyzed (Participants) | 7
  Month 90: Markedly Improved | 0 [0.0 to 41.0]
  Month 90: Moderately Improved: number analyzed (Participants) | 7
  Month 90: Moderately Improved | 0 [0.0 to 41.0]
  Month 90: Mildly Improved: number analyzed (Participants) | 7
  Month 90: Mildly Improved | 42.9 [9.9 to 81.6]
  Month 90: Unchanged: number analyzed (Participants) | 7
  Month 90: Unchanged | 28.6 [3.7 to 71.0]
  Month 90: Mildly Worsened: number analyzed (Participants) | 7
  Month 90: Mildly Worsened | 28.6 [3.7 to 71.0]
  Month 90: Moderately Worsened: number analyzed (Participants) | 7
  Month 90: Moderately Worsened | 0 [0.0 to 41.0]
  Month 90: Markedly Worsened: number analyzed (Participants) | 7
  Month 90: Markedly Worsened | 0 [0.0 to 41.0]
  Month 96: Markedly Improved: number analyzed (Participants) | 4
  Month 96: Markedly Improved | 0 [0.0 to 60.2]
  Month 96: Moderately Improved: number analyzed (Participants) | 4
  Month 96: Moderately Improved | 0 [0.0 to 60.2]
  Month 96: Mildly Improved: number analyzed (Participants) | 4
  Month 96: Mildly Improved | 0 [0.0 to 60.2]
  Month 96: Unchanged: number analyzed (Participants) | 4
  Month 96: Unchanged | 25.0 [0.6 to 80.6]
  Month 96: Mildly Worsened: number analyzed (Participants) | 4
  Month 96: Mildly Worsened | 50.0 [6.8 to 93.2]
  Month 96: Moderately Worsened: number analyzed (Participants) | 4
  Month 96: Moderately Worsened | 25.0 [0.6 to 80.6]
  Month 96: Markedly Worsened: number analyzed (Participants) | 4
  Month 96: Markedly Worsened | 0 [0.0 to 60.2]
  Month 102: Markedly Improved: number analyzed (Participants) | 4
  Month 102: Markedly Improved | 0 [0.0 to 60.2]
  Month 102: Moderately Improved: number analyzed (Participants) | 4
  Month 102: Moderately Improved | 0 [0.0 to 60.2]
  Month 102: Mildly Improved: number analyzed (Participants) | 4
  Month 102: Mildly Improved | 0 [0.0 to 60.2]
  Month 102: Unchanged: number analyzed (Participants) | 4
  Month 102: Unchanged | 75.0 [19.4 to 99.4]
  Month 102: Mildly Worsened: number analyzed (Participants) | 4
  Month 102: Mildly Worsened | 0 [0.0 to 60.2]
  Month 102: Moderately Worsened: number analyzed (Participants) | 4
  Month 102: Moderately Worsened | 0 [0.0 to 60.2]
  Month 102: Markedly Worsened: number analyzed (Participants) | 4
  Month 102: Markedly Worsened | 25.0 [0.6 to 80.6]
  Month 108: Markedly Improved: number analyzed (Participants) | 5
  Month 108: Markedly Improved | 40.0 [5.3 to 85.3]
  Month 108: Moderately Improved: number analyzed (Participants) | 5
  Month 108: Moderately Improved | 0 [0.0 to 52.2]
  Month 108: Mildly Improved: number analyzed (Participants) | 5
  Month 108: Mildly Improved | 20.0 [0.5 to 71.6]
  Month 108: Unchanged: number analyzed (Participants) | 5
  Month 108: Unchanged | 40.0 [5.3 to 85.3]
  Month 108: Mildly Worsened: number analyzed (Participants) | 5
  Month 108: Mildly Worsened | 0 [0.0 to 52.2]
  Month 108: Moderately Worsened: number analyzed (Participants) | 5
  Month 108: Moderately Worsened | 0 [0.0 to 52.2]
  Month 108: Markedly Worsened: number analyzed (Participants) | 5
  Month 108: Markedly Worsened | 0 [0.0 to 52.2]
  Month 114: Markedly Improved: number analyzed (Participants) | 4
  Month 114: Markedly Improved | 0 [0.0 to 60.2]
  Month 114: Moderately Improved: number analyzed (Participants) | 4
  Month 114: Moderately Improved | 0 [0.0 to 60.2]
  Month 114: Mildly Improved: number analyzed (Participants) | 4
  Month 114: Mildly Improved | 25.0 [0.6 to 80.6]
  Month 114: Unchanged: number analyzed (Participants) | 4
  Month 114: Unchanged | 0 [0.0 to 60.2]
  Month 114: Mildly Worsened: number analyzed (Participants) | 4
  Month 114: Mildly Worsened | 75.0 [19.4 to 99.4]
  Month 114: Moderately Worsened: number analyzed (Participants) | 4
  Month 114: Moderately Worsened | 0 [0.0 to 60.2]
  Month 114: Markedly Worsened: number analyzed (Participants) | 4
  Month 114: Markedly Worsened | 0 [0.0 to 60.2]
  Month 120: Markedly Improved: number analyzed (Participants) | 2
  Month 120: Markedly Improved | 0 [0.0 to 84.2]
  Month 120: Moderately Improved: number analyzed (Participants) | 2
  Month 120: Moderately Improved | 0 [0.0 to 84.2]
  Month 120: Mildly Improved: number analyzed (Participants) | 2
  Month 120: Mildly Improved | 50.0 [1.3 to 98.7]
  Month 120: Unchanged: number analyzed (Participants) | 2
  Month 120: Unchanged | 50.0 [1.3 to 98.7]
  Month 120: Mildly Worsened: number analyzed (Participants) | 2
  Month 120: Mildly Worsened | 0 [0.0 to 84.2]
  Month 120: Moderately Worsened: number analyzed (Participants) | 2
  Month 120: Moderately Worsened | 0 [0.0 to 84.2]
  Month 120: Markedly Worsened: number analyzed (Participants) | 2
  Month 120: Markedly Worsened | 0 [0.0 to 84.2]
  Month 126: Markedly Improved: number analyzed (Participants) | 2
  Month 126: Markedly Improved | 0 [0.0 to 84.2]
  Month 126: Moderately Improved: number analyzed (Participants) | 2
  Month 126: Moderately Improved | 0 [0.0 to 84.2]
  Month 126: Mildly Improved: number analyzed (Participants) | 2
  Month 126: Mildly Improved | 0 [0.0 to 84.2]
  Month 126: Unchanged: number analyzed (Participants) | 2
  Month 126: Unchanged | 0 [0.0 to 84.2]
  Month 126: Mildly Worsened: number analyzed (Participants) | 2
  Month 126: Mildly Worsened | 100.0 [15.8 to 100.0]
  Month 126: Moderately Worsened: number analyzed (Participants) | 2
  Month 126: Moderately Worsened | 0 [0.0 to 84.2]
  Month 126: Markedly Worsened: number analyzed (Participants) | 2
  Month 126: Markedly Worsened | 0 [0.0 to 84.2]
  Month 132: Markedly Improved: number analyzed (Participants) | 1
  Month 132: Markedly Improved | 0 [0.0 to 97.5]
  Month 132: Moderately Improved: number analyzed (Participants) | 1
  Month 132: Moderately Improved | 0 [0.0 to 97.5]
  Month 132: Mildly Improved: number analyzed (Participants) | 1
  Month 132: Mildly Improved | 0 [0.0 to 97.5]
  Month 132: Unchanged: number analyzed (Participants) | 1
  Month 132: Unchanged | 0 [0.0 to 97.5]
  Month 132: Mildly Worsened: number analyzed (Participants) | 1
  Month 132: Mildly Worsened | 100.0 [2.5 to 100.0]
  Month 132: Moderately Worsened: number analyzed (Participants) | 1
  Month 132: Moderately Worsened | 0 [0.0 to 97.5]
  Month 132: Markedly Worsened: number analyzed (Participants) | 1
  Month 132: Markedly Worsened | 0 [0.0 to 97.5]

21. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Classification at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126 and 132
Description: as for outcome 4
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126, 132
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants
  Month 6: Worsened | 5
  Month 6: Unchanged | 25
  Month 6: Improved | 1
  Month 18: Worsened: number analyzed (Participants) | 27
  Month 18: Worsened | 7
  Month 18: Unchanged: number analyzed (Participants) | 27
  Month 18: Unchanged | 17
  Month 18: Improved: number analyzed (Participants) | 27
  Month 18: Improved | 3
  Month 24: Worsened: number analyzed (Participants) | 22
  Month 24: Worsened | 7
  Month 24: Unchanged: number analyzed (Participants) | 22
  Month 24: Unchanged | 12
  Month 24: Improved: number analyzed (Participants) | 22
  Month 24: Improved | 3
  Month 30: Worsened: number analyzed (Participants) | 20
  Month 30: Worsened | 4
  Month 30: Unchanged: number analyzed (Participants) | 20
  Month 30: Unchanged | 14
  Month 30: Improved: number analyzed (Participants) | 20
  Month 30: Improved | 2
  Month 36: Worsened: number analyzed (Participants) | 19
  Month 36: Worsened | 6
  Month 36: Unchanged: number analyzed (Participants) | 19
  Month 36: Unchanged | 11
  Month 36: Improved: number analyzed (Participants) | 19
  Month 36: Improved | 2
  Month 42: Worsened: number analyzed (Participants) | 17
  Month 42: Worsened | 10
  Month 42: Unchanged: number analyzed (Participants) | 17
  Month 42: Unchanged | 5
  Month 42: Improved: number analyzed (Participants) | 17
  Month 42: Improved | 2
  Month 48: Worsened: number analyzed (Participants) | 12
  Month 48: Worsened | 6
  Month 48: Unchanged: number analyzed (Participants) | 12
  Month 48: Unchanged | 4
  Month 48: Improved: number analyzed (Participants) | 12
  Month 48: Improved | 2
  Month 54: Worsened: number analyzed (Participants) | 12
  Month 54: Worsened | 6
  Month 54: Unchanged: number analyzed (Participants) | 12
  Month 54: Unchanged | 6
  Month 54: Improved: number analyzed (Participants) | 12
  Month 54: Improved | 0
  Month 66: Worsened: number analyzed (Participants) | 6
  Month 66: Worsened | 5
  Month 66: Unchanged: number analyzed (Participants) | 6
  Month 66: Unchanged | 1
  Month 66: Improved: number analyzed (Participants) | 6
  Month 66: Improved | 0
  Month 72: Worsened: number analyzed (Participants) | 7
  Month 72: Worsened | 2
  Month 72: Unchanged: number analyzed (Participants) | 7
  Month 72: Unchanged | 5
  Month 72: Improved: number analyzed (Participants) | 7
  Month 72: Improved | 0
  Month 78: Worsened: number analyzed (Participants) | 7
  Month 78: Worsened | 3
  Month 78: Unchanged: number analyzed (Participants) | 7
  Month 78: Unchanged | 4
  Month 78: Improved: number analyzed (Participants) | 7
  Month 78: Improved | 0
  Month 84: Worsened: number analyzed (Participants) | 6
  Month 84: Worsened | 3
  Month 84: Unchanged: number analyzed (Participants) | 6
  Month 84: Unchanged | 3
  Month 84: Improved: number analyzed (Participants) | 6
  Month 84: Improved | 0
  Month 90: Worsened: number analyzed (Participants) | 7
  Month 90: Worsened | 3
  Month 90: Unchanged: number analyzed (Participants) | 7
  Month 90: Unchanged | 4
  Month 90: Improved: number analyzed (Participants) | 7
  Month 90: Improved | 0
  Month 96: Worsened: number analyzed (Participants) | 5
  Month 96: Worsened | 3
  Month 96: Unchanged: number analyzed (Participants) | 5
  Month 96: Unchanged | 1
  Month 96: Improved: number analyzed (Participants) | 5
  Month 96: Improved | 1
  Month 102: Worsened: number analyzed (Participants) | 5
  Month 102: Worsened | 2
  Month 102: Unchanged: number analyzed (Participants) | 5
  Month 102: Unchanged | 2
  Month 102: Improved: number analyzed (Participants) | 5
  Month 102: Improved | 1
  Month 108: Worsened: number analyzed (Participants) | 5
  Month 108: Worsened | 2
  Month 108: Unchanged: number analyzed (Participants) | 5
  Month 108: Unchanged | 1
  Month 108: Improved: number analyzed (Participants) | 5
  Month 108: Improved | 2
  Month 114: Worsened: number analyzed (Participants) | 4
  Month 114: Worsened | 2
  Month 114: Unchanged: number analyzed (Participants) | 4
  Month 114: Unchanged | 2
  Month 114: Improved: number analyzed (Participants) | 4
  Month 114: Improved | 0
  Month 120: Worsened: number analyzed (Participants) | 4
  Month 120: Worsened | 3
  Month 120: Unchanged: number analyzed (Participants) | 4
  Month 120: Unchanged | 1
  Month 120: Improved: number analyzed (Participants) | 4
  Month 120: Improved | 0
  Month 126: Worsened: number analyzed (Participants) | 2
  Month 126: Worsened | 1
  Month 126: Unchanged: number analyzed (Participants) | 2
  Month 126: Unchanged | 1
  Month 126: Improved: number analyzed (Participants) | 2
  Month 126: Improved | 0
  Month 132: Worsened: number analyzed (Participants) | 1
  Month 132: Worsened | 1
  Month 132: Unchanged: number analyzed (Participants) | 1
  Month 132: Unchanged | 0
  Month 132: Improved: number analyzed (Participants) | 1
  Month 132: Improved | 0

22. Secondary Outcome: Change From Baseline in Total Distance Walked During 6 Minute Walk Test (6MWT) at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120 and 132
Description: as for outcome 6
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 132
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
meters
  Change at Month 6 | 2.9 (60.64)
  Change at Month 18: number analyzed (Participants) | 21
  Change at Month 18 | -21.6 (108.19)
  Change at Month 24: number analyzed (Participants) | 20
  Change at Month 24 | -15.7 (78.39)
  Change at Month 30: number analyzed (Participants) | 18
  Change at Month 30 | -44.5 (111.67)
  Change at Month 36: number analyzed (Participants) | 17
  Change at Month 36 | -63.5 (101.37)
  Change at Month 42: number analyzed (Participants) | 16
  Change at Month 42 | -95.2 (124.79)
  Change at Month 48: number analyzed (Participants) | 11
  Change at Month 48 | -110.9 (128.57)
  Change at Month 54: number analyzed (Participants) | 11
  Change at Month 54 | -127.8 (124.01)
  Change at Month 66: number analyzed (Participants) | 4
  Change at Month 66 | -63.2 (114.20)
  Change at Month 72: number analyzed (Participants) | 3
  Change at Month 72 | -139.5 (210.18)
  Change at Month 78: number analyzed (Participants) | 3
  Change at Month 78 | -94.3 (177.01)
  Change at Month 84: number analyzed (Participants) | 4
  Change at Month 84 | -100.3 (151.71)
  Change at Month 90: number analyzed (Participants) | 6
  Change at Month 90 | -97.6 (125.50)
  Change at Month 96: number analyzed (Participants) | 4
  Change at Month 96 | -118.9 (114.20)
  Change at Month 102: number analyzed (Participants) | 3
  Change at Month 102 | -82.3 (19.30)
  Change at Month 108: number analyzed (Participants) | 5
  Change at Month 108 | -141.9 (112.29)
  Change at Month 114: number analyzed (Participants) | 4
  Change at Month 114 | -166.9 (137.23)
  Change at Month 120: number analyzed (Participants) | 3
  Change at Month 120 | -184.5 (82.22)
  Change at Month 132: number analyzed (Participants) | 1
  Change at Month 132 | -289.6

23. Secondary Outcome: Number of Participants Categorized Based on Total Distance Walked During 6 Minute Walk Test (6MWT) at Baseline, Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126 and 132
Description: as for outcome 9
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126, 132
Population: ITT population included all participants who were enrolled and received at least 1 dose of study medication, had baseline and at least 1 post-baseline cardiac measure. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure. "Number analyzed" =participants evaluable for this outcome measure at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 30
Participants
  Baseline: Level 1 | 8
  Baseline: Level 2 | 10
  Baseline: Level 3 | 7
  Baseline: Level 4 | 5
  Month 6: Level 1 | 7
  Month 6: Level 2 | 9
  Month 6: Level 3 | 9
  Month 6: Level 4 | 5
  Month 18:Level 1: number analyzed (Participants) | 21
  Month 18:Level 1 | 5
  Month 18: Level 2: number analyzed (Participants) | 21
  Month 18: Level 2 | 5
  Month 18: Level 3: number analyzed (Participants) | 21
  Month 18: Level 3 | 8
  Month 18: Level 4: number analyzed (Participants) | 21
  Month 18: Level 4 | 3
  Month 24: Level 1: number analyzed (Participants) | 20
  Month 24: Level 1 | 3
  Month 24: Level 2: number analyzed (Participants) | 20
  Month 24: Level 2 | 7
  Month 24: Level 3: number analyzed (Participants) | 20
  Month 24: Level 3 | 4
  Month 24: Level 4: number analyzed (Participants) | 20
  Month 24: Level 4 | 6
  Month 30: Level 1: number analyzed (Participants) | 18
  Month 30: Level 1 | 5
  Month 30: Level 2: number analyzed (Participants) | 18
  Month 30: Level 2 | 6
  Month 30: Level 3: number analyzed (Participants) | 18
  Month 30: Level 3 | 6
  Month 30: Level 4: number analyzed (Participants) | 18
  Month 30: Level 4 | 1
  Month 36: Level 1: number analyzed (Participants) | 17
  Month 36: Level 1 | 5
  Month 36: Level 2: number analyzed (Participants) | 17
  Month 36: Level 2 | 4
  Month 36: Level 3: number analyzed (Participants) | 17
  Month 36: Level 3 | 6
  Month 36: Level 4: number analyzed (Participants) | 17
  Month 36: Level 4 | 2
  Month 42: Level 1: number analyzed (Participants) | 16
  Month 42: Level 1 | 9
  Month 42: Level 2: number analyzed (Participants) | 16
  Month 42: Level 2 | 2
  Month 42: Level 3: number analyzed (Participants) | 16
  Month 42: Level 3 | 4
  Month 42: Level 4: number analyzed (Participants) | 16
  Month 42: Level 4 | 1
  Month 48: Level 1: number analyzed (Participants) | 11
  Month 48: Level 1 | 5
  Month 48: Level 2: number analyzed (Participants) | 11
  Month 48: Level 2 | 1
  Month 48: Level 3: number analyzed (Participants) | 11
  Month 48: Level 3 | 5
  Month 48: Level 4: number analyzed (Participants) | 11
  Month 48: Level 4 | 0
  Month 54: Level 1: number analyzed (Participants) | 11
  Month 54: Level 1 | 7
  Month 54: Level 2: number analyzed (Participants) | 11
  Month 54: Level 2 | 2
  Month 54: Level 3: number analyzed (Participants) | 11
  Month 54: Level 3 | 1
  Month 54: Level 4: number analyzed (Participants) | 11
  Month 54: Level 4 | 1
  Month 66: Level 1: number analyzed (Participants) | 4
  Month 66: Level 1 | 2
  Month 66: Level 2: number analyzed (Participants) | 4
  Month 66: Level 2 | 1
  Month 66: Level 3: number analyzed (Participants) | 4
  Month 66: Level 3 | 1
  Month 66: Level 4: number analyzed (Participants) | 4
  Month 66: Level 4 | 0
  Month 72: Level 1: number analyzed (Participants) | 3
  Month 72: Level 1 | 2
  Month 72: Level 2: number analyzed (Participants) | 3
  Month 72: Level 2 | 0
  Month 72: Level 3: number analyzed (Participants) | 3
  Month 72: Level 3 | 1
  Month 72: Level 4: number analyzed (Participants) | 3
  Month 72: Level 4 | 0
  Month 78: Level 1: number analyzed (Participants) | 3
  Month 78: Level 1 | 2
  Month 78: Level 2: number analyzed (Participants) | 3
  Month 78: Level 2 | 0
  Month 78: Level 3: number analyzed (Participants) | 3
  Month 78: Level 3 | 1
  Month 78: Level 4: number analyzed (Participants) | 3
  Month 78: Level 4 | 0
  Month 84: Level 1: number analyzed (Participants) | 4
  Month 84: Level 1 | 2
  Month 84: Level 2: number analyzed (Participants) | 4
  Month 84: Level 2 | 2
  Month 84: Level 3: number analyzed (Participants) | 4
  Month 84: Level 3 | 0
  Month 84: Level 4: number analyzed (Participants) | 4
  Month 84: Level 4 | 0
  Month 90: Level 1: number analyzed (Participants) | 6
  Month 90: Level 1 | 3
  Month 90: Level 2: number analyzed (Participants) | 6
  Month 90: Level 2 | 1
  Month 90: Level 3: number analyzed (Participants) | 6
  Month 90: Level 3 | 2
  Month 90: Level 4: number analyzed (Participants) | 6
  Month 90: Level 4 | 0
  Month 96: Level 1: number analyzed (Participants) | 4
  Month 96: Level 1 | 3
  Month 96: Level 2: number analyzed (Participants) | 4
  Month 96: Level 2 | 1
  Month 96: Level 3: number analyzed (Participants) | 4
  Month 96: Level 3 | 0
  Month 96: Level 4: number analyzed (Participants) | 4
  Month 96: Level 4 | 0
  Month 102: Level 1: number analyzed (Participants) | 3
  Month 102: Level 1 | 0
  Month 102: Level 2: number analyzed (Participants) | 3
  Month 102: Level 2 | 2
  Month 102: Level 3: number analyzed (Participants) | 3
  Month 102: Level 3 | 1
  Month 102: Level 4: number analyzed (Participants) | 3
  Month 102: Level 4 | 0
  Month 108: Level 1: number analyzed (Participants) | 5
  Month 108: Level 1 | 3
  Month 108: Level 2: number analyzed (Participants) | 5
  Month 108: Level 2 | 2
  Month 108: Level 3: number analyzed (Participants) | 5
  Month 108: Level 3 | 0
  Month 108: Level 4: number analyzed (Participants) | 5
  Month 108: Level 4 | 0
  Month 114: Level 1: number analyzed (Participants) | 4
  Month 114: Level 1 | 3
  Month 114: Level 2: number analyzed (Participants) | 4
  Month 114: Level 2 | 1
  Month 114: Level 3: number analyzed (Participants) | 4
  Month 114: Level 3 | 0
  Month 114: Level 4: number analyzed (Participants) | 4
  Month 114: Level 4 | 0
  Month 120: Level 1: number analyzed (Participants) | 3
  Month 120: Level 1 | 1
  Month 120: Level 2: number analyzed (Participants) | 3
  Month 120: Level 2 | 2
  Month 120: Level 3: number analyzed (Participants) | 3
  Month 120: Level 3 | 0
  Month 120: Level 4: number analyzed (Participants) | 3
  Month 120: Level 4 | 0
  Month 132: Level 1: number analyzed (Participants) | 1
  Month 132: Level 1 | 1
  Month 132: Level 2: number analyzed (Participants) | 1
  Month 132: Level 2 | 0
  Month 132: Level 3: number analyzed (Participants) | 1
  Month 132: Level 3 | 0
  Month 132: Level 4: number analyzed (Participants) | 1
  Month 132: Level 4 | 0

24. Secondary Outcome: Change From Baseline in Dyspnea and Fatigue Scores During 6 Minute Walk Test (6MWT) at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120 and 132
Description: 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. Participants were asked to walk as far as possible for 6 minutes at a pace that was comfortable to them, and were permitted to slow down, to stop, and to rest as necessary. Dyspnea: participants were asked to rate the difficulty of their breathing, pre-walk and post-walk at each visit, on a scale of range 0 (no breathlessness at all) to 10 (maximum breathlessness). Higher scores indicated more severity. Fatigue: participants were asked to rate the how tired they felt, pre-walk and post-walk at each visit, on a scale of range 0 (not at all) to 10 (maximal) Higher scores indicated more fatigue. At each visit, scores for pre-walk test, post-walk test and within visit difference (difference from post-walk to pre-walk) were evaluated. Change from baseline was calculated for each pre-walk test, post-walk test and within visit difference at specified visits.
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 132
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 28
units on a scale
  Dyspnea: Change at Month 6, Pre walk | 0.3 (1.32)
  Dyspnea: Change at Month 6, Post walk | 0.9 (1.54)
  Dyspnea: Change at Month 6,Within Visit Difference | 0.6 (1.56)
  Dyspnea: Change at Month 18, Pre walk: number analyzed (Participants) | 19
  Dyspnea: Change at Month 18, Pre walk | 0.3 (1.11)
  Dyspnea: Change at Month 18, Post walk: number analyzed (Participants) | 19
  Dyspnea: Change at Month 18, Post walk | 0.8 (1.40)
  Dyspnea:Change at Month 18,Within Visit Difference: number analyzed (Participants) | 19
  Dyspnea:Change at Month 18,Within Visit Difference | 0.6 (1.93)
  Dyspnea: Change at Month 24, Pre walk: number analyzed (Participants) | 18
  Dyspnea: Change at Month 24, Pre walk | 0.3 (0.75)
  Dyspnea: Change at Month 24, Post walk: number analyzed (Participants) | 18
  Dyspnea: Change at Month 24, Post walk | 1.5 (1.91)
  Dyspnea:Change at Month 24,Within Visit Difference: number analyzed (Participants) | 18
  Dyspnea:Change at Month 24,Within Visit Difference | 1.1 (2.02)
  Dyspnea: Change at Month 30, Pre walk: number analyzed (Participants) | 17
  Dyspnea: Change at Month 30, Pre walk | 0.2 (0.47)
  Dyspnea: Change at Month 30, Post walk: number analyzed (Participants) | 17
  Dyspnea: Change at Month 30, Post walk | 1.2 (1.27)
  Dyspnea:Change at Month 30,Within Visit Difference: number analyzed (Participants) | 17
  Dyspnea:Change at Month 30,Within Visit Difference | 1.0 (1.36)
  Dyspnea: Change at Month 36, Pre walk: number analyzed (Participants) | 16
  Dyspnea: Change at Month 36, Pre walk | 0.1 (1.36)
  Dyspnea: Change at Month 36, Post walk: number analyzed (Participants) | 16
  Dyspnea: Change at Month 36, Post walk | -0.2 (2.68)
  Dyspnea:Change at Month 36,Within Visit Difference: number analyzed (Participants) | 16
  Dyspnea:Change at Month 36,Within Visit Difference | -0.3 (1.97)
  Dyspnea: Change at Month 42, Pre walk: number analyzed (Participants) | 15
  Dyspnea: Change at Month 42, Pre walk | 0.5 (0.90)
  Dyspnea: Change at Month 42, Post walk: number analyzed (Participants) | 15
  Dyspnea: Change at Month 42, Post walk | 1.0 (1.45)
  Dyspnea:Change at Month 42,Within Visit Difference: number analyzed (Participants) | 15
  Dyspnea:Change at Month 42,Within Visit Difference | 0.5 (1.53)
  Dyspnea: Change at Month 48, Pre walk: number analyzed (Participants) | 10
  Dyspnea: Change at Month 48, Pre walk | 0.6 (1.17)
  Dyspnea: Change at Month 48, Post walk: number analyzed (Participants) | 10
  Dyspnea: Change at Month 48, Post walk | 1.3 (0.98)
  Dyspnea:Change at Month 48,Within Visit Difference: number analyzed (Participants) | 10
  Dyspnea:Change at Month 48,Within Visit Difference | 0.8 (1.64)
  Dyspnea: Change at Month 54, Pre walk: number analyzed (Participants) | 11
  Dyspnea: Change at Month 54, Pre walk | 0.4 (1.56)
  Dyspnea: Change at Month 54, Post walk: number analyzed (Participants) | 10
  Dyspnea: Change at Month 54, Post walk | 1.0 (1.93)
  Dyspnea:Change at Month 54,Within Visit Difference: number analyzed (Participants) | 10
  Dyspnea:Change at Month 54,Within Visit Difference | 0.6 (1.91)
  Dyspnea: Change at Month 66, Pre walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 66, Pre walk | 1.4 (1.11)
  Dyspnea: Change at Month 66, Post walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 66, Post walk | 1.5 (1.29)
  Dyspnea:Change at Month 66,Within Visit Difference: number analyzed (Participants) | 4
  Dyspnea:Change at Month 66,Within Visit Difference | 0.1 (1.18)
  Dyspnea: Change at Month 72, Pre walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 72, Pre walk | 0.8 (1.44)
  Dyspnea: Change at Month 72, Post walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 72, Post walk | 0.7 (1.15)
  Dyspnea:Change at Month 72,Within Visit Difference: number analyzed (Participants) | 3
  Dyspnea:Change at Month 72,Within Visit Difference | -0.2 (0.29)
  Dyspnea: Change at Month 78, Pre walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 78, Pre walk | 2.2 (2.02)
  Dyspnea: Change at Month 78, Post walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 78, Post walk | 0.7 (0.58)
  Dyspnea:Change at Month 78,Within Visit Difference: number analyzed (Participants) | 3
  Dyspnea:Change at Month 78,Within Visit Difference | -1.5 (1.50)
  Dyspnea: Change at Month 84, Pre walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 84, Pre walk | -0.1 (0.85)
  Dyspnea: Change at Month 84, Post walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 84, Post walk | 0.5 (1.00)
  Dyspnea:Change at Month 84,Within Visit Difference: number analyzed (Participants) | 4
  Dyspnea:Change at Month 84,Within Visit Difference | 0.6 (1.70)
  Dyspnea: Change at Month 90, Pre walk: number analyzed (Participants) | 6
  Dyspnea: Change at Month 90, Pre walk | 0.6 (0.66)
  Dyspnea: Change at Month 90, Post walk: number analyzed (Participants) | 6
  Dyspnea: Change at Month 90, Post walk | -0.8 (2.32)
  Dyspnea:Change at Month 90,Within Visit Difference: number analyzed (Participants) | 6
  Dyspnea:Change at Month 90,Within Visit Difference | -1.4 (2.20)
  Dyspnea: Change at Month 96, Pre walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 96, Pre walk | 1.0 (1.41)
  Dyspnea: Change at Month 96, Post walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 96, Post walk | 1.3 (1.50)
  Dyspnea:Change at Month 96,Within Visit Difference: number analyzed (Participants) | 4
  Dyspnea:Change at Month 96,Within Visit Difference | 0.3 (2.36)
  Dyspnea: Change at Month 102, Pre walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 102, Pre walk | -0.3 (0.58)
  Dyspnea: Change at Month 102, Post walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 102, Post walk | -1.3 (4.04)
  Dyspnea:Change at Month102,Within Visit Difference: number analyzed (Participants) | 3
  Dyspnea:Change at Month102,Within Visit Difference | -1.0 (3.46)
  Dyspnea: Change at Month 108, Pre walk: number analyzed (Participants) | 5
  Dyspnea: Change at Month 108, Pre walk | 1.7 (2.82)
  Dyspnea: Change at Month 108, Post walk: number analyzed (Participants) | 5
  Dyspnea: Change at Month 108, Post walk | 0.7 (4.97)
  Dyspnea:Change at Month108,Within Visit Difference: number analyzed (Participants) | 5
  Dyspnea:Change at Month108,Within Visit Difference | -1.0 (2.81)
  Dyspnea: Change at Month 114, Pre walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 114, Pre walk | 0.4 (1.80)
  Dyspnea: Change at Month 114, Post walk: number analyzed (Participants) | 4
  Dyspnea: Change at Month 114, Post walk | 0.1 (0.63)
  Dyspnea:Change at Month114,Within Visit Difference: number analyzed (Participants) | 4
  Dyspnea:Change at Month114,Within Visit Difference | -0.3 (1.19)
  Dyspnea: Change at Month 120, Pre walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 120, Pre walk | 0.3 (1.53)
  Dyspnea: Change at Month 120, Post walk: number analyzed (Participants) | 3
  Dyspnea: Change at Month 120, Post walk | -0.8 (1.04)
  Dyspnea:Change at Month120,Within Visit Difference: number analyzed (Participants) | 3
  Dyspnea:Change at Month120,Within Visit Difference | -1.2 (2.47)
  Dyspnea: Change at Month 132, Pre walk: number analyzed (Participants) | 1
  Dyspnea: Change at Month 132, Pre walk | -1.0
  Dyspnea: Change at Month 132, Post walk: number analyzed (Participants) | 1
  Dyspnea: Change at Month 132, Post walk | -1.0
  Dyspnea:Change at Month132,Within Visit Difference: number analyzed (Participants) | 1
  Dyspnea:Change at Month132,Within Visit Difference | 0.0
  Fatigue: Change at Month 6, Pre walk | 0.2 (1.69)
  Fatigue: Change at Month 6, Post walk | 0.7 (2.82)
  Fatigue:Change at Month 6,Within Visit Difference | 0.4 (2.92)
  Fatigue: Change at Month 18, Pre walk: number analyzed (Participants) | 19
  Fatigue: Change at Month 18, Pre walk | 0.0 (2.13)
  Fatigue: Change at Month 18, Post walk: number analyzed (Participants) | 19
  Fatigue: Change at Month 18, Post walk | 0.2 (1.40)
  Fatigue:Change at Month 18,Within Visit Difference: number analyzed (Participants) | 19
  Fatigue:Change at Month 18,Within Visit Difference | 0.2 (2.51)
  Fatigue: Change at Month 24, Pre walk: number analyzed (Participants) | 18
  Fatigue: Change at Month 24, Pre walk | 0.1 (1.66)
  Fatigue: Change at Month 24, Post walk: number analyzed (Participants) | 18
  Fatigue: Change at Month 24, Post walk | 1.0 (2.33)
  Fatigue:Change at Month 24,Within Visit Difference: number analyzed (Participants) | 18
  Fatigue:Change at Month 24,Within Visit Difference | 0.9 (2.97)
  Fatigue: Change at Month 30, Pre walk: number analyzed (Participants) | 17
  Fatigue: Change at Month 30, Pre walk | -0.4 (1.58)
  Fatigue: Change at Month 30, Post walk: number analyzed (Participants) | 17
  Fatigue: Change at Month 30, Post walk | 0.9 (1.65)
  Fatigue:Change at Month 30,Within Visit Difference: number analyzed (Participants) | 17
  Fatigue:Change at Month 30,Within Visit Difference | 1.3 (2.23)
  Fatigue: Change at Month 36, Pre walk: number analyzed (Participants) | 16
  Fatigue: Change at Month 36, Pre walk | -0.2 (2.29)
  Fatigue: Change at Month 36, Post walk: number analyzed (Participants) | 16
  Fatigue: Change at Month 36, Post walk | 0.8 (2.05)
  Fatigue:Change at Month 36,Within Visit Difference: number analyzed (Participants) | 16
  Fatigue:Change at Month 36,Within Visit Difference | 1.0 (2.76)
  Fatigue: Change at Month 42, Pre walk: number analyzed (Participants) | 15
  Fatigue: Change at Month 42, Pre walk | 0.4 (1.76)
  Fatigue: Change at Month 42, Post walk: number analyzed (Participants) | 15
  Fatigue: Change at Month 42, Post walk | 1.6 (1.86)
  Fatigue:Change at Month 42,Within Visit Difference: number analyzed (Participants) | 15
  Fatigue:Change at Month 42,Within Visit Difference | 1.2 (2.86)
  Fatigue: Change at Month 48, Pre walk: number analyzed (Participants) | 10
  Fatigue: Change at Month 48, Pre walk | 0.6 (1.26)
  Fatigue: Change at Month 48, Post walk: number analyzed (Participants) | 10
  Fatigue: Change at Month 48, Post walk | 1.5 (1.84)
  Fatigue:Change at Month 48,Within Visit Difference: number analyzed (Participants) | 10
  Fatigue:Change at Month 48,Within Visit Difference | 0.9 (2.38)
  Fatigue: Change at Month 54, Pre walk: number analyzed (Participants) | 11
  Fatigue: Change at Month 54, Pre walk | 0.5 (1.57)
  Fatigue: Change at Month 54, Post walk: number analyzed (Participants) | 10
  Fatigue: Change at Month 54, Post walk | 0.5 (1.90)
  Fatigue:Change at Month 54,Within Visit Difference: number analyzed (Participants) | 10
  Fatigue:Change at Month 54,Within Visit Difference | -0.1 (1.97)
  Fatigue: Change at Month 66, Pre walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 66, Pre walk | 0.3 (0.50)
  Fatigue: Change at Month 66, Post walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 66, Post walk | 0.5 (2.38)
  Fatigue:Change at Month 66,Within Visit Difference: number analyzed (Participants) | 4
  Fatigue:Change at Month 66,Within Visit Difference | 0.3 (2.22)
  Fatigue: Change at Month 72, Pre walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 72, Pre walk | 2.0 (1.73)
  Fatigue: Change at Month 72, Post walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 72, Post walk | 1.0 (1.73)
  Fatigue:Change at Month 72,Within Visit Difference: number analyzed (Participants) | 3
  Fatigue:Change at Month 72,Within Visit Difference | -1.0 (0.00)
  Fatigue: Change at Month 78, Pre walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 78, Pre walk | 2.0 (2.00)
  Fatigue: Change at Month 78, Post walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 78, Post walk | 1.0 (2.65)
  Fatigue:Change at Month 78,Within Visit Difference: number analyzed (Participants) | 3
  Fatigue:Change at Month 78,Within Visit Difference | -1.0 (1.00)
  Fatigue: Change at Month 84, Pre walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 84, Pre walk | 0.0 (0.82)
  Fatigue: Change at Month 84, Post walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 84, Post walk | 0.4 (1.11)
  Fatigue:Change at Month 84,Within Visit Difference: number analyzed (Participants) | 4
  Fatigue:Change at Month 84,Within Visit Difference | 0.4 (1.49)
  Fatigue: Change at Month 90, Pre walk: number analyzed (Participants) | 6
  Fatigue: Change at Month 90, Pre walk | 1.3 (1.75)
  Fatigue: Change at Month 90, Post walk: number analyzed (Participants) | 6
  Fatigue: Change at Month 90, Post walk | -0.3 (2.07)
  Fatigue:Change at Month 90,Within Visit Difference: number analyzed (Participants) | 6
  Fatigue:Change at Month 90,Within Visit Difference | -1.7 (3.27)
  Fatigue: Change at Month 96, Pre walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 96, Pre walk | 0.8 (1.50)
  Fatigue: Change at Month 96, Post walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 96, Post walk | 0.0 (0.82)
  Fatigue:Change at Month 96,Within Visit Difference: number analyzed (Participants) | 4
  Fatigue:Change at Month 96,Within Visit Difference | -0.8 (1.71)
  Fatigue: Change at Month 102, Pre walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 102, Pre walk | 1.0 (2.65)
  Fatigue: Change at Month 102, Post walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 102, Post walk | -0.7 (1.53)
  Fatigue:Change at Month102,Within Visit Difference: number analyzed (Participants) | 3
  Fatigue:Change at Month102,Within Visit Difference | -1.7 (1.15)
  Fatigue: Change at Month 108, Pre walk: number analyzed (Participants) | 5
  Fatigue: Change at Month 108, Pre walk | 1.8 (2.77)
  Fatigue: Change at Month 108, Post walk: number analyzed (Participants) | 5
  Fatigue: Change at Month 108, Post walk | 0.9 (3.54)
  Fatigue:Change at Month108,Within Visit Difference: number analyzed (Participants) | 5
  Fatigue:Change at Month108,Within Visit Difference | -0.9 (1.14)
  Fatigue: Change at Month 114, Pre walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 114, Pre walk | 1.0 (2.16)
  Fatigue: Change at Month 114, Post walk: number analyzed (Participants) | 4
  Fatigue: Change at Month 114, Post walk | -0.1 (0.85)
  Fatigue:Change at Month114,Within Visit Difference: number analyzed (Participants) | 4
  Fatigue:Change at Month114,Within Visit Difference | -1.1 (1.44)
  Fatigue: Change at Month 120, Pre walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 120, Pre walk | 0.0 (1.00)
  Fatigue: Change at Month 120, Post walk: number analyzed (Participants) | 3
  Fatigue: Change at Month 120, Post walk | -1.2 (0.76)
  Fatigue:Change at Month120,Within Visit Difference: number analyzed (Participants) | 3
  Fatigue:Change at Month120,Within Visit Difference | -1.2 (1.76)
  Fatigue: Change at Month 132, Pre walk: number analyzed (Participants) | 1
  Fatigue: Change at Month 132, Pre walk | -1.0
  Fatigue: Change at Month 132, Post walk: number analyzed (Participants) | 1
  Fatigue: Change at Month 132, Post walk | -0.5
  Fatigue:Change at Month132,Within Visit Difference: number analyzed (Participants) | 1
  Fatigue:Change at Month132,Within Visit Difference | 0.5

25. Secondary Outcome: Number of Participants Categorized on Basis of Change From Baseline in Total Distance Walked During 6 Minute Walk Test (6MWT) at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120 and 132
Description: as for outcome 12
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 132
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 30
Participants
  Month 6: Worsened | 5
  Month 6: Unchanged | 20
  Month 6: Improved | 5
  Month 18: Worsened: number analyzed (Participants) | 21
  Month 18: Worsened | 9
  Month 18: Unchanged: number analyzed (Participants) | 21
  Month 18: Unchanged | 7
  Month 18: Improved: number analyzed (Participants) | 21
  Month 18: Improved | 5
  Month 24: Worsened: number analyzed (Participants) | 20
  Month 24: Worsened | 6
  Month 24: Unchanged: number analyzed (Participants) | 20
  Month 24: Unchanged | 10
  Month 24: Improved: number analyzed (Participants) | 20
  Month 24: Improved | 4
  Month 30: Worsened: number analyzed (Participants) | 18
  Month 30: Worsened | 9
  Month 30: Unchanged: number analyzed (Participants) | 18
  Month 30: Unchanged | 4
  Month 30: Improved: number analyzed (Participants) | 18
  Month 30: Improved | 5
  Month 36: Worsened: number analyzed (Participants) | 17
  Month 36: Worsened | 8
  Month 36: Unchanged: number analyzed (Participants) | 17
  Month 36: Unchanged | 7
  Month 36: Improved: number analyzed (Participants) | 17
  Month 36: Improved | 2
  Month 42: Worsened: number analyzed (Participants) | 16
  Month 42: Worsened | 9
  Month 42: Unchanged: number analyzed (Participants) | 16
  Month 42: Unchanged | 6
  Month 42: Improved: number analyzed (Participants) | 16
  Month 42: Improved | 1
  Month 48: Worsened: number analyzed (Participants) | 11
  Month 48: Worsened | 7
  Month 48: Unchanged: number analyzed (Participants) | 11
  Month 48: Unchanged | 3
  Month 48: Improved: number analyzed (Participants) | 11
  Month 48: Improved | 1
  Month 54: Worsened: number analyzed (Participants) | 11
  Month 54: Worsened | 7
  Month 54: Unchanged: number analyzed (Participants) | 11
  Month 54: Unchanged | 4
  Month 54: Improved: number analyzed (Participants) | 11
  Month 54: Improved | 0
  Month 66: Worsened: number analyzed (Participants) | 4
  Month 66: Worsened | 3
  Month 66: Unchanged: number analyzed (Participants) | 4
  Month 66: Unchanged | 1
  Month 66: Improved: number analyzed (Participants) | 4
  Month 66: Improved | 0
  Month 72: Worsened: number analyzed (Participants) | 3
  Month 72: Worsened | 2
  Month 72: Unchanged: number analyzed (Participants) | 3
  Month 72: Unchanged | 1
  Month 72: Improved: number analyzed (Participants) | 3
  Month 72: Improved | 0
  Month 78: Worsened: number analyzed (Participants) | 3
  Month 78: Worsened | 2
  Month 78: Unchanged: number analyzed (Participants) | 3
  Month 78: Unchanged | 1
  Month 78: Improved: number analyzed (Participants) | 3
  Month 78: Improved | 0
  Month 84: Worsened: number analyzed (Participants) | 4
  Month 84: Worsened | 3
  Month 84: Unchanged: number analyzed (Participants) | 4
  Month 84: Unchanged | 1
  Month 84: Improved: number analyzed (Participants) | 4
  Month 84: Improved | 0
  Month 90: Worsened: number analyzed (Participants) | 6
  Month 90: Worsened | 4
  Month 90: Unchanged: number analyzed (Participants) | 6
  Month 90: Unchanged | 1
  Month 90: Improved: number analyzed (Participants) | 6
  Month 90: Improved | 1
  Month 96: Worsened: number analyzed (Participants) | 4
  Month 96: Worsened | 3
  Month 96: Unchanged: number analyzed (Participants) | 4
  Month 96: Unchanged | 1
  Month 96: Improved: number analyzed (Participants) | 4
  Month 96: Improved | 0
  Month 102: Worsened: number analyzed (Participants) | 3
  Month 102: Worsened | 2
  Month 102: Unchanged: number analyzed (Participants) | 3
  Month 102: Unchanged | 1
  Month 102: Improved: number analyzed (Participants) | 3
  Month 102: Improved | 0
  Month 108: Worsened: number analyzed (Participants) | 5
  Month 108: Worsened | 4
  Month 108: Unchanged: number analyzed (Participants) | 5
  Month 108: Unchanged | 1
  Month 108: Improved: number analyzed (Participants) | 5
  Month 108: Improved | 0
  Month 114: Worsened: number analyzed (Participants) | 4
  Month 114: Worsened | 3
  Month 114: Unchanged: number analyzed (Participants) | 4
  Month 114: Unchanged | 1
  Month 114: Improved: number analyzed (Participants) | 4
  Month 114: Improved | 0
  Month 120: Worsened: number analyzed (Participants) | 3
  Month 120: Worsened | 3
  Month 120: Unchanged: number analyzed (Participants) | 3
  Month 120: Unchanged | 0
  Month 120: Improved: number analyzed (Participants) | 3
  Month 120: Improved | 0
  Month 132: Worsened: number analyzed (Participants) | 1
  Month 132: Worsened | 1
  Month 132: Unchanged: number analyzed (Participants) | 1
  Month 132: Unchanged | 0
  Month 132: Improved: number analyzed (Participants) | 1
  Month 132: Improved | 0

26. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Summary Score at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126 and 132
Description: as for outcome 14
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126, 132
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
units on a scale
  Overall Summary Score: Change at Month 6 | -2.12 (12.423)
  Overall Summary Score: Change at Month 18: number analyzed (Participants) | 28
  Overall Summary Score: Change at Month 18 | -4.58 (18.926)
  Overall Summary Score: Change at Month 24: number analyzed (Participants) | 22
  Overall Summary Score: Change at Month 24 | -2.94 (16.247)
  Overall Summary Score: Change at Month 30: number analyzed (Participants) | 20
  Overall Summary Score: Change at Month 30 | -5.41 (17.695)
  Overall Summary Score: Change at Month 36: number analyzed (Participants) | 19
  Overall Summary Score: Change at Month 36 | -6.86 (18.525)
  Overall Summary Score: Change at Month 42: number analyzed (Participants) | 17
  Overall Summary Score: Change at Month 42 | -12.76 (23.646)
  Overall Summary Score: Change at Month 48: number analyzed (Participants) | 12
  Overall Summary Score: Change at Month 48 | -13.22 (24.893)
  Overall Summary Score: Change at Month 54: number analyzed (Participants) | 13
  Overall Summary Score: Change at Month 54 | -14.99 (23.688)
  Overall Summary Score: Change at Month 66: number analyzed (Participants) | 6
  Overall Summary Score: Change at Month 66 | -1.77 (30.476)
  Overall Summary Score: Change at Month 72: number analyzed (Participants) | 7
  Overall Summary Score: Change at Month 72 | 0.41 (23.317)
  Overall Summary Score: Change at Month 78: number analyzed (Participants) | 7
  Overall Summary Score: Change at Month 78 | -3.60 (24.231)
  Overall Summary Score: Change at Month 84: number analyzed (Participants) | 6
  Overall Summary Score: Change at Month 84 | -3.72 (32.770)
  Overall Summary Score: Change at Month 90: number analyzed (Participants) | 7
  Overall Summary Score: Change at Month 90 | -0.28 (30.296)
  Overall Summary Score: Change at Month 96: number analyzed (Participants) | 4
  Overall Summary Score: Change at Month 96 | -17.84 (47.842)
  Overall Summary Score: Change at Month 102: number analyzed (Participants) | 4
  Overall Summary Score: Change at Month 102 | -12.63 (40.904)
  Overall Summary Score: Change at Month 108: number analyzed (Participants) | 4
  Overall Summary Score: Change at Month 108 | -1.19 (35.375)
  Overall Summary Score: Change at Month 114: number analyzed (Participants) | 4
  Overall Summary Score: Change at Month 114 | -2.99 (37.897)
  Overall Summary Score: Change at Month 120: number analyzed (Participants) | 2
  Overall Summary Score: Change at Month 120 | -35.55 (9.023)
  Overall Summary Score: Change at Month 126: number analyzed (Participants) | 2
  Overall Summary Score: Change at Month 126 | -39.32 (8.102)
  Overall Summary Score: Change at Month 132: number analyzed (Participants) | 1
  Overall Summary Score: Change at Month 132 | -40.10
  Clinical Summary Score: Change at Month 6 | -3.00 (11.650)
  Clinical Summary Score: Change at Month 18: number analyzed (Participants) | 28
  Clinical Summary Score: Change at Month 18 | -6.66 (17.340)
  Clinical Summary Score: Change at Month 24: number analyzed (Participants) | 22
  Clinical Summary Score: Change at Month 24 | -2.87 (15.875)
  Clinical Summary Score: Change at Month 30: number analyzed (Participants) | 20
  Clinical Summary Score: Change at Month 30 | -7.80 (17.497)
  Clinical Summary Score: Change at Month 36: number analyzed (Participants) | 19
  Clinical Summary Score: Change at Month 36 | -9.53 (17.700)
  Clinical Summary Score: Change at Month 42: number analyzed (Participants) | 17
  Clinical Summary Score: Change at Month 42 | -17.05 (22.804)
  Clinical Summary Score: Change at Month 48: number analyzed (Participants) | 12
  Clinical Summary Score: Change at Month 48 | -15.67 (24.854)
  Clinical Summary Score: Change at Month 54: number analyzed (Participants) | 13
  Clinical Summary Score: Change at Month 54 | -16.90 (21.295)
  Clinical Summary Score: Change at Month 66: number analyzed (Participants) | 6
  Clinical Summary Score: Change at Month 66 | -3.45 (27.219)
  Clinical Summary Score: Change at Month 72: number analyzed (Participants) | 7
  Clinical Summary Score: Change at Month 72 | -1.82 (21.558)
  Clinical Summary Score: Change at Month 78: number analyzed (Participants) | 7
  Clinical Summary Score: Change at Month 78 | -7.13 (22.422)
  Clinical Summary Score: Change at Month 84: number analyzed (Participants) | 6
  Clinical Summary Score: Change at Month 84 | -6.53 (29.881)
  Clinical Summary Score: Change at Month 90: number analyzed (Participants) | 7
  Clinical Summary Score: Change at Month 90 | -2.47 (24.198)
  Clinical Summary Score: Change at Month 96: number analyzed (Participants) | 4
  Clinical Summary Score: Change at Month 96 | -19.27 (42.768)
  Clinical Summary Score: Change at Month 102: number analyzed (Participants) | 4
  Clinical Summary Score: Change at Month 102 | -15.10 (31.690)
  Clinical Summary Score: Change at Month 108: number analyzed (Participants) | 4
  Clinical Summary Score: Change at Month 108 | -3.26 (27.764)
  Clinical Summary Score: Change at Month 114: number analyzed (Participants) | 4
  Clinical Summary Score: Change at Month 114 | -4.69 (32.213)
  Clinical Summary Score: Change at Month 120: number analyzed (Participants) | 2
  Clinical Summary Score: Change at Month 120 | -42.45 (11.417)
  Clinical Summary Score: Change at Month 126: number analyzed (Participants) | 2
  Clinical Summary Score: Change at Month 126 | -38.02 (14.731)
  Clinical Summary Score: Change at Month 132: number analyzed (Participants) | 1
  Clinical Summary Score: Change at Month 132 | -40.63

27. Secondary Outcome: Number of Participants With Abnormalities in Echocardiography
Description: Echocardiography abnormalities included: absent respiratory variation of inferior vena cava, any valve thickening, aortic valve thickening, decreased respiratory variation of inferior vena cava, dilated inferior vena cava, E deceleration time less than or equal to (<=) 150 millisecond, E wave/A Wave (E/A) ratio >=2, ejection fraction < 50%, isovolumic relaxation time (IVRT) <=70 millisecond, left ventricular posterior wall thickness >=13 millimeter (mm), left ventricular septal thickness >= 13 mm, mitral valve thickening, pericardial effusion, pulmonary valve thickening, right ventricular thickness >=7 mm, tricuspid valve thickening, ratio between early mitral inflow velocity and mitral annular early diastolic velocity (e/e') Lateral greater than (>) 15, e/e' Septal >15.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants | 31

28. Secondary Outcome: Change From Baseline in Troponin I and Troponin T Serum Levels at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120 and 126
Description: as for outcome 16
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120 and 126
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
nanogram per milliliter
  Troponin I: Change at Month 6 | -0.016 (0.0533)
  Troponin I: Change at Month 18: number analyzed (Participants) | 27
  Troponin I: Change at Month 18 | 0.032 (0.1307)
  Troponin I: Change at Month 24: number analyzed (Participants) | 22
  Troponin I: Change at Month 24 | 0.023 (0.0986)
  Troponin I: Change at Month 30: number analyzed (Participants) | 20
  Troponin I: Change at Month 30 | 0.022 (0.1038)
  Troponin I: Change at Month 36: number analyzed (Participants) | 19
  Troponin I: Change at Month 36 | 0.029 (0.1099)
  Troponin I: Change at Month 42: number analyzed (Participants) | 17
  Troponin I: Change at Month 42 | 0.042 (0.1409)
  Troponin I: Change at Month 48: number analyzed (Participants) | 12
  Troponin I: Change at Month 48 | 0.058 (0.1409)
  Troponin I: Change at Month 54: number analyzed (Participants) | 13
  Troponin I: Change at Month 54 | 0.042 (0.1226)
  Troponin I: Change at Month 66: number analyzed (Participants) | 6
  Troponin I: Change at Month 66 | -0.012 (0.0133)
  Troponin I: Change at Month 72: number analyzed (Participants) | 4
  Troponin I: Change at Month 72 | -0.010 (0.0183)
  Troponin I: Change at Month 78: number analyzed (Participants) | 3
  Troponin I: Change at Month 78 | -0.013 (0.0208)
  Troponin I: Change at Month 84: number analyzed (Participants) | 4
  Troponin I: Change at Month 84 | -0.008 (0.0096)
  Troponin I: Change at Month 90: number analyzed (Participants) | 7
  Troponin I: Change at Month 90 | -0.003 (0.0293)
  Troponin I: Change at Month 96: number analyzed (Participants) | 4
  Troponin I: Change at Month 96 | -0.008 (0.0150)
  Troponin I: Change at Month 102: number analyzed (Participants) | 4
  Troponin I: Change at Month 102 | -0.010 (0.0356)
  Troponin I: Change at Month 108: number analyzed (Participants) | 5
  Troponin I: Change at Month 108 | 0.000 (0.0071)
  Troponin I: Change at Month 114: number analyzed (Participants) | 4
  Troponin I: Change at Month 114 | 0.000 (0.0271)
  Troponin I: Change at Month 120: number analyzed (Participants) | 2
  Troponin I: Change at Month 120 | 0.000 (0.0141)
  Troponin I: Change at Month 126: number analyzed (Participants) | 2
  Troponin I: Change at Month 126 | 0.005 (0.0354)
  Troponin T: Change at Month 6: number analyzed (Participants) | 29
  Troponin T: Change at Month 6 | -0.0007 (0.01710)
  Troponin T: Change at Month 18: number analyzed (Participants) | 27
  Troponin T: Change at Month 18 | 0.0271 (0.07429)
  Troponin T: Change at Month 24: number analyzed (Participants) | 22
  Troponin T: Change at Month 24 | 0.0132 (0.03286)
  Troponin T: Change at Month 30: number analyzed (Participants) | 20
  Troponin T: Change at Month 30 | 0.0166 (0.02227)
  Troponin T: Change at Month 36: number analyzed (Participants) | 19
  Troponin T: Change at Month 36 | 0.0205 (0.03049)
  Troponin T: Change at Month 42: number analyzed (Participants) | 17
  Troponin T: Change at Month 42 | 0.0329 (0.05665)
  Troponin T: Change at Month 48: number analyzed (Participants) | 10
  Troponin T: Change at Month 48 | 0.0510 (0.09562)
  Troponin T: Change at Month 54: number analyzed (Participants) | 13
  Troponin T: Change at Month 54 | 0.0562 (0.13264)
  Troponin T: Change at Month 66: number analyzed (Participants) | 6
  Troponin T: Change at Month 66 | 0.0050 (0.02588)
  Troponin T: Change at Month 72: number analyzed (Participants) | 4
  Troponin T: Change at Month 72 | -0.0055 (0.01714)
  Troponin T: Change at Month 78: number analyzed (Participants) | 3
  Troponin T: Change at Month 78 | 0.0000 (0.01732)
  Troponin T: Change at Month 84: number analyzed (Participants) | 4
  Troponin T: Change at Month 84 | -0.0003 (0.01415)
  Troponin T: Change at Month 90: number analyzed (Participants) | 7
  Troponin T: Change at Month 90 | 0.0026 (0.00962)
  Troponin T: Change at Month 96: number analyzed (Participants) | 3
  Troponin T: Change at Month 96 | -0.0037 (0.00551)
  Troponin T: Change at Month 102: number analyzed (Participants) | 4
  Troponin T: Change at Month 102 | 0.0098 (0.01461)
  Troponin T: Change at Month 108: number analyzed (Participants) | 5
  Troponin T: Change at Month 108 | 0.0100 (0.00707)
  Troponin T: Change at Month114: number analyzed (Participants) | 4
  Troponin T: Change at Month114 | 0.0100 (0.00816)
  Troponin T: Change at Month 120: number analyzed (Participants) | 2
  Troponin T: Change at Month 120 | 0.0150 (0.02121)
  Troponin T: Change at Month 126: number analyzed (Participants) | 1
  Troponin T: Change at Month 126 | 0.0000

29. Secondary Outcome: Change From Baseline in Amino-Terminal B-type Natriuretic Peptide (NT-proBNP) Serum Level at Months 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120 and 126
Description: NT-proBNP was biomarker of cardiac stress (myocardial necrosis and increased filling pressures/ LV wall stress).
Time Frame: Baseline, Month 6, 18, 24, 30, 36, 42, 48, 54, 66, 72, 78, 84, 90, 96, 102, 108, 114, 120, 126
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
nanogram per milliliter
  Change at Month 6 | 66.0 (2164.66)
  Change at Month 18: number analyzed (Participants) | 27
  Change at Month 18 | 492.0 (2455.65)
  Change at Month 24: number analyzed (Participants) | 22
  Change at Month 24 | 211.5 (2119.01)
  Change at Month 30: number analyzed (Participants) | 20
  Change at Month 30 | 701.8 (2423.16)
  Change at Month 36: number analyzed (Participants) | 19
  Change at Month 36 | 1063.5 (2813.85)
  Change at Month 42: number analyzed (Participants) | 17
  Change at Month 42 | 2510.2 (5143.47)
  Change at Month 48: number analyzed (Participants) | 10
  Change at Month 48 | 3761.2 (7892.80)
  Change at Month 54: number analyzed (Participants) | 12
  Change at Month 54 | 1668.1 (2677.27)
  Change at Month 66: number analyzed (Participants) | 6
  Change at Month 66 | 433.3 (493.76)
  Change at Month 72: number analyzed (Participants) | 4
  Change at Month 72 | 625.5 (471.41)
  Change at Month 78: number analyzed (Participants) | 3
  Change at Month 78 | 707.7 (236.53)
  Change at Month 84: number analyzed (Participants) | 4
  Change at Month 84 | 348.5 (700.98)
  Change at Month 90: number analyzed (Participants) | 7
  Change at Month 90 | 283.7 (971.53)
  Change at Month 96: number analyzed (Participants) | 3
  Change at Month 96 | 1453.0 (2193.75)
  Change at Month 102: number analyzed (Participants) | 4
  Change at Month 102 | 1439.0 (2032.43)
  Change at Month 108: number analyzed (Participants) | 5
  Change at Month 108 | 346.4 (1279.58)
  Change at Month 114: number analyzed (Participants) | 3
  Change at Month 114 | 465.7 (790.48)
  Change at Month 120: number analyzed (Participants) | 2
  Change at Month 120 | 1232.0 (667.51)
  Change at Month 126: number analyzed (Participants) | 1
  Change at Month 126 | 1249.0

30. Secondary Outcome: Number of Participants With All-cause Hospitalization and Cardiac-related Hospitalization Events
Description: All cause hospitalization was defined as any serious adverse event, which resulted in hospitalization. Cardiac-related hospitalization was any hospitalization meeting the following criteria: cardiac disorders or AE preferred term as chest discomfort, chest pain, death, cerebrovascular accident, embolic stroke, disease progression.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants
  All-cause Hospitalization | 27
  Cardiac Related Hospitalization | 18

31. Secondary Outcome: Time to All-cause Mortality and Cardiac-Related Mortality
Description: Time to death for all participants with a death date in Clinical Database, or censored at the last dose date + 28 days for those participants who were alive at the end of the study is reported.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
years
  All-Cause Mortality | 4.1 [1.9 to 5.4]
  Cardiac-related mortality | 5.9 [3.0 to NA] — Due to very less number of events upper limit of 95% CI could not be estimated, hence not provided.

32. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and all non-serious adverse events.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants
  Participants with AEs | 31
  Participants with SAEs | 29

33. Secondary Outcome: Number of Participants With Treatment-Related Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and all non-serious adverse events. Relatedness to study drug was assessed by the investigator as (Yes/No).
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants
  Participant with AEs | 7
  Participant with SAEs | 4

34. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included examination of general appearance, endocrine, head and neck, cardiovascular, eyes, abdomen, ears, skin, nose, musculoskeletal, throat, neurological, respiratory, immunologic/allergies, genitourinary, hematologic/lymphatic. Clinical significance of any physical examination finding was judged by investigator.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: Safety analysis population included all participants who were enrolled in this study and who had taken at least 1 dose of study medication. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 28
Participants | 19

35. Secondary Outcome: Number of Participants With Any Concomitant Medications
Description: Number of participants who used medication other than study drug were reported.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants | 31

36. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval (millisecond), RR interval (millisecond), QRS interval (millisecond), QT and QTc interval (millisecond) and heart rate (beats per minute). Clinical significance of any ECG finding was judged by investigator.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants | 1

37. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory parameters included hematology and biochemistry: alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen, gamma glutamyl transferase (GGT), creatinine, total bilirubin, international normalized ratio (INR), troponin I, troponin T, prothrombin time, sodium, globulin potassium, chloride, bicarbonate, cholesterol, calcium, uric acid, inorganic phosphorous, thyroid-stimulating hormone, glucose, total thyroxine (T4), free T4, total proteins, prealbumin (transthyretin), albumin, hemoglobin, platelets, hematocrit, white blood cell count, red blood cell count, neutrophils, packed cell volume, lymphocytes, mean corpuscular volume, monocytes, mean corpuscular hemoglobin, eosinophils, mean corpuscular hemoglobin concentration, basophils, retinol-binding protein, Urinalysis: bilirubin, pH, blood (free Hb), protein, nitrite, glucose, urobilinogen, ketones, specific gravity.
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tafamidis 20 mg
Number analyzed (Participants) | 31
Participants | 27

ADVERSE EVENTS:
Time Frame: Post-Month 12 up to Month 132 (approximately 10 years) of Study FX1B-303
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population evaluated.
Arm/Group | Tafamidis 20 mg
All-Cause Mortality (participants affected / at risk) | 23/31
Serious Adverse Events (participants affected / at risk) | 29/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg (N=31)
Anaemia (Blood and lymphatic system disorders) | 1
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
ATRIAL FLUTTER (Cardiac disorders) | 1
ATRIAL TACHYCARDIA (Cardiac disorders) | 2
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1
CARDIAC AMYLOIDOSIS (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 6
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 9
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
FAMILIAL AMYLOIDOSIS (Congenital, familial and genetic disorders) | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
FAECALOMA (Gastrointestinal disorders) | 2
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
OESOPHAGEAL MOTILITY DISORDER (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
ASTHENIA (General disorders) | 2
CHEST DISCOMFORT (General disorders) | 2
CHEST PAIN (General disorders) | 3
DEATH (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
BACTERIAL SEPSIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 3
DEVICE RELATED INFECTION (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 2
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
SEPSIS (Infections and infestations) | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1
UROSEPSIS (Infections and infestations) | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1
CARDIAC CONTUSION (Injury, poisoning and procedural complications) | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 6
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
SKIN LACERATION (Injury, poisoning and procedural complications) | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
WEIGHT INCREASED (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1
GOUT (Metabolism and nutrition disorders) | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DEMENTIA (Nervous system disorders) | 1
EMBOLIC STROKE (Nervous system disorders) | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1
PARKINSONISM (Nervous system disorders) | 1
PRESYNCOPE (Nervous system disorders) | 2
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
HALLUCINATION (Psychiatric disorders) | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2
END STAGE RENAL DISEASE (Renal and urinary disorders) | 1
POLYURIA (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 2
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1
VARICOSE VEIN RUPTURED (Vascular disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis 20 mg (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 5
CARDIAC FAILURE (Cardiac disorders) | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3
PALPITATIONS (Cardiac disorders) | 3
FAMILIAL AMYLOIDOSIS (Congenital, familial and genetic disorders) | 2
HYPOTHYROIDISM (Endocrine disorders) | 3
CATARACT (Eye disorders) | 3
ATRIAL FLUTTER (Cardiac disorders) | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 11
DIARRHOEA (Gastrointestinal disorders) | 5
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 3
ASTHENIA (General disorders) | 4
CHEST PAIN (General disorders) | 2
GAIT DISTURBANCE (General disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 5
PERIPHERAL SWELLING (General disorders) | 2
PYREXIA (General disorders) | 3
BRONCHITIS (Infections and infestations) | 3
CELLULITIS (Infections and infestations) | 3
EAR INFECTION (Infections and infestations) | 2
NASOPHARYNGITIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 4
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5
URINARY TRACT INFECTION (Infections and infestations) | 6
CONTUSION (Injury, poisoning and procedural complications) | 4
FALL (Injury, poisoning and procedural complications) | 13
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2
RIB FRACTURE (Injury, poisoning and procedural complications) | 2
SKIN ABRASION (Injury, poisoning and procedural complications) | 3
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 2
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 2
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 3
PROTHROMBIN TIME PROLONGED (Investigations) | 2
VENOUS PRESSURE JUGULAR INCREASED (Investigations) | 2
WEIGHT DECREASED (Investigations) | 6
WEIGHT INCREASED (Investigations) | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 7
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 3
FLUID OVERLOAD (Metabolism and nutrition disorders) | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
BALANCE DISORDER (Nervous system disorders) | 5
DIZZINESS (Nervous system disorders) | 5
DIZZINESS POSTURAL (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 3
MEMORY IMPAIRMENT (Nervous system disorders) | 2
SYNCOPE (Nervous system disorders) | 3
TREMOR (Nervous system disorders) | 3
DEPRESSION (Psychiatric disorders) | 3
MENTAL STATUS CHANGES (Psychiatric disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 2
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 4
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3
URTICARIA (Skin and subcutaneous tissue disorders) | 2
HYPOTENSION (Vascular disorders) | 4
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2
FATIGUE (General disorders) | 10
SKIN LACERATION (Injury, poisoning and procedural complications) | 7
INSOMNIA (Psychiatric disorders) | 3
HAEMATURIA (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2012-06-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT00935012/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT00935012/SAP_001.pdf